CLINICAL TRIAL: NCT02897544
Title: Developing a Health Education Intervention for Breast Cancer Survivorship
Brief Title: Integrative Approaches for Cancer Survivorship 2: Project 2
Acronym: IACS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-1856
Record Dates: First submitted 2016-09-07; First posted 2016-09-13 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Health Education Intervention (Experimental): Study participants will attend Health Education sessions led by health educators over the course of 6 months. The emphasis in the sessions will be to provide engaging educational information on common survivorship issues.
  Interventions: Behavioral: Individualized Manualized Health Education Intervention

INTERVENTIONS:
Behavioral: Individualized Manualized Health Education Intervention

SUMMARY:
The purpose of this study is to develop and test a 6 month manualized Health Education intervention in recent breast cancer survivors.

DETAILED DESCRIPTION:
Post-treatment cancer survivorship is often associated with a void in care given the drop-off in support provided to survivors from the medical team as well as family and friends. The investigators aim to develop and test a Health Education intervention in breast cancer survivors. Specifically, the investigators aim to develop the manualized Health Education intervention; to assess feasibility; and to provide preliminary data on the effects of the intervention. The data from this pilot study will be used to inform future study.

ELIGIBILITY:
Inclusion Criteria:

* Female breast cancer survivor who is over 1 month and less than 24 months beyond the completion of primary therapy (surgery, radiation, and chemotherapy)
* Having received chemotherapy as part of their primary therapy for breast cancer
* Be in complete remission
* Aged 18 years or older
* Able to read, write, and understand English
* Karnofsky Performance Status (KPS) greater than or equal to 60
* Have impaired quality of life
* Ability to give informed consent

Exclusion Criteria:

* Receiving chemotherapy or radiotherapy at the time of study enrollment. Anti-her2 directed therapy is not exclusionary.
* Being within 1 month (before or after) of surgery for breast cancer (including breast reconstructive surgery). Smaller surgical procedures such as implant exchange are not exclusionary.
* Patients on adjuvant hormone therapy for less than 2 months
* Have surgery for breast cancer or breast reconstructive surgery planned during the initial 6 month study period. Smaller surgical procedures such as implant exchange are not exclusionary.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Change in quality of life over 6 months | Baseline, 3 months, 6 months
  The investigators will use the EORTC QLQ C30 in conjunction with a breast cancer-specific subscale, BR23, to collect data on quality of life and cancer-related symptoms.

SECONDARY OUTCOMES:
Change in fatigue over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Lee Fatigue Scale (LFS) to collect data on fatigue.
Change in sleep quality over 6 months | Baseline, 3 months, 6 months
  The investigators will use the General Sleep Disturbance Scale (GSDS) to collect data on sleep disturbance.
Change in anxiety over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Spielberger State Anxiety Inventory (STAI-S) to collect data on anxiety.
Change in depressive symptoms over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Center for Epidemiological Studies - Depression Scale (CES-D) to collect data on depressive symptoms.
Change in pain over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Brief Pain Inventory (BPI) to collect data on pain intensity and interference with function.
Change in diet over 6 months | Baseline, 3 months, 6 months
  The investigators will use the Automated Self-Administered 24-hour Recall (ASA24) to assess dietary recall over a 24 hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Dhruva, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Osher Center for Integrative Medicine, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No